CLINICAL TRIAL: NCT02292238
Title: Benfotiamine in Alzheimer's Disease: A Pilot Study
Acronym: Benfotiamine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Collaborators: Burke Rehabilitation Hospital (Other); Columbia University (Other); National Institute on Aging (NIA) (NIH); Alzheimer's Drug Discovery Foundation (Other); Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Gary E. Gibson, Professor of Neuroscience; Brain and Mind Institute; Weill Cornell Med College, Burke Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRC-451; 1R01AG043679-01A1 (NIH)
Record Dates: First submitted 2014-11-10; First posted 2014-11-17 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; benfotiamine; glucose; Amyloid
MeSH Terms: conditions — Alzheimer Disease | interventions — benphothiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Benfotiamine (Experimental): The patients in this arm will be treated with benfotiamine
  Interventions: Drug: Benfotiamine
- Placebo (Placebo Comparator): The patients in this arm will be treated with placebo
  Interventions: Drug: Benfotiamine

INTERVENTIONS:
Drug: Benfotiamine — * To test whether increasing brain thiamine by administering 600 mg per day (300 mg/morning and 300 mg/evening) of benfotiamine for one year can slow cognitive decline in these patients as measured with the Alzheimer's Disease Assessment Scale (ADAS-COG).
  * To determine whether increasing brain thiamine availability with 600 mg (300 mg/morning and 300 mg/evening) per day of benfotiamine for one year can slow the decline in brain glucose metabolism in these patients as measured with Fluorodeoxyglucose Positron Emission Tomography(FGPET) in the posterior cingulate.
  Other Names: S-[2-{[(4-amino-2- methylpyrimidin-5-yl)methyl] (formyl)amino}-5-(phosphonooxy)pent-2-en-3-yl] benzenecarbothioate

SUMMARY:
General Investigational Plan

Study Objectives The goal of this proposal is to determine whether enhancing brain glucose utilization minimizes cognitive decline in patients with Amnestic Mild Cognitive Impairment (AMCI) or mild Alzheimer's disease (AD) dementia. We propose a proof of concept double-blind, placebo controlled pilot study to determine if increasing brain thiamine availability with the investigational new drug benfotiamine, will minimize the decline in glucose utilization and slow the cognitive decline associated with the progression AMCI/AD dementia.

Specifically, our objectives are two-fold:

* To test whether increasing brain thiamine by administering 600 mg per day (300 mg/morning and 300 mg/evening) of benfotiamine for one year can slow cognitive decline in these patients as measured with the Alzheimer's Disease Assessment Scale (ADAS-COG).
* To determine whether increasing brain thiamine availability with 600 mg (300 mg/morning and 300 mg/evening) per day of benfotiamine for one year can slow the decline in brain glucose metabolism in these patients as measured with Fluorodeoxyglucose Positron Emission Tomography(FGPET) in the posterior cingulate.

We will also carry out the following secondary objectives:

* Assess if there are differences in secondary clinical outcome measures (NPI, ADCSADL, CDR, Buschke) between benfotiamine and placebo groups and whether specific cognitive domains (ie: activities of daily living, learning and memory verbal memory, behavioral, etc.) are driving these changes.
* Compare ADAS-COG change scores in the benfotiamine and placebo groups within and between strata that were defined by initial cognitive impairment, to attempt to identified the population that most benefits from benfotiamine.
* Compare changes in glucose utilization between the benfotiamine and placebo groups in secondary Regions of Interest (ROIs) including the hippocampus, prefrontal regions and entorhinal cortex.
* Compare changes in whole brain glucose utilization between the benfotiamine and placebo groups using statistical parametric mapping (SPM).
* Assess the correlation between changes in glucose utilization with changes in ADAS Cog.
* Determine if ApoE4 genotype alters the response to benfotiamine.

DETAILED DESCRIPTION:
Study Design

This study will be conducted at the Burke Rehabilitation Hospital under an IRB protocol. Wplan to accrue a total of 76 male and/or female patients (> 65 years) with a diagnosis of AMCI/AD dementia that are also amyloid positive by PET scan. Patients will be randomized and blinded to either a benfotiamine or placebo group. Because it is unknown whether there will be differential responses to treatment according to initial cognitive impairment, participants will be stratified according to the median MMSE cut-off score of our historical METS population who are > 65 years old and have an MMSE >21.

In this double-blind study, patients and their caregivers, as well as all physicians, clinicians, coordinators and investigators interacting with the patients, will be unaware of the treatment assignments. Treatment assignments will be available to the safety-monitoring physician, Dr. Michael Reding, who will have no unnecessary subject contact. If necessary, the code will be revealed to Dr. Reding by the pharmacist, Dr. Thomas Grandville.

Each patient will make six visits to the Memory Evaluation and Treatment Service (METS) clinic at Burke Rehabilitation Hospital. Information on medication use, vital signs, outcome measures, compliance and safety/tolerability will be collected at each time point. The screening visit (visit 1) will take place within 30 days prior to baseline visit (visit 2). Informed consent/assent will be obtained from each subject or his/her caregiver prior to conducting any study related procedures. During the screening visit a review of inclusion/exclusion criteria will be completed along with the collection of demographic data, disease history, and information about prior and concomitant medications. A complete medical history, physical examination, neurological examination, including the MMSE, CDR, CSDD and vital signs, will be collected. Blood will be drawn to assess blood glucose Patients that are diagnosed as likely Alzheimer patients that are not hyperglycemic will then have an amyloid PET scan. Only patients with a diagnosis of AD and a positive amyloid scan will be included. Prior to baseline (visit 2), FDGPET studies will be completed for each subject. At the baseline visit (visit 2) blood will be drawn to determine APOE and thiamine (vitamin B1 status). At visits 2-6, information on concomitant medications will be updated, vitals will be taken, medication compliance will be assessed and the following study measures will be administered: Alzheimer's Disease Assessment Scale (ADASCog), Buschke SRT, Neuropsychological Inventory (NPI), Clinical Dementia Rating Scale (CDR) and Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADLs). The final PET scan will be conducted approximately one week prior to the last visit. In addition to safety assessments at time of each visit, each patient will receive a call from the clinical coordinator at weeks 2 and 6 to assess for adverse events.

The benfotiamine and placebo will be dispensed by the pharmacy at Burke under the direction of Thomas Grandville, D. Pharm. The caregiver will administer the drug since patients with memory problems may forget to take it on a regular basis. In the placebo group, the active compound benfotiamine will be replaced with microcrystalline cellulose. The other components, shape and color are identical to the treatment. Caregivers will be instructed to oversee the administration of the study medication as prescribed to ensure compliance. A record of the number of capsules dispensed, number returned, and actual number taken will be recorded at scheduled visits. Each patient will be treated for 12 months.

The study cognitive measures include: the ADAS-Cog (our primary outcome measure), Alzheimer's Disease Cooperative Study-Activities of Daily Living, Neuropsychiatric Inventory, Clinical Dementia Rating Scale, Buschke Selective Reminding Test (SRT). is a standard diagnostic tool in the assessment of verbal memory. The Biological/Mechanistic Outcome Measures will be FDG-PET Scanning Procedures

Data Analysis Preliminary analyses will be conducted to describe the study sample and to confirm the relationship between level of glucose utilization and severity of cognitive impairment. For continuous variables (eg cognitive function, glucose utilization), we will first examine distributions to assess normality assumptions. We will perform transformations as needed to stabilize the variance, and to reduce skewness and kurtosis. We will use means (sd) and proportions n (%) to characterize the study sample. T-tests and Chi-square, or Wilcoxon rank sum test and Fisher, where appropriate, will be used to assess for any differences in patient characteristics according to treatment group. We will use spearman correlation coefficients and linear regression, unadjusted and adjusted for covariates, to assess the relationship between FDG-PET and MMSE in the whole population as well as in MMSE stratified groups to examine the relationship between initial MMSE score and glucose uptake.

All analyses to test study hypotheses will be run as intention to treat (ITT). Missing observations will be addressed by using the method of last observation carried forward (LOCF).

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Clinical diagnosis of AMCI by the Peterson criteria or probable AD dementia according to the National Institute of Neurological Disorders and stroke and the Alzheimer's Disease related Disorders Association (NINCDS/ADRDA)
* MMSE score > or equal to 21
* CDR score > or equal to 0.5 and < or equal to1
* Cornell Scale for Depression in Dementia(CSDD) score <10.
* Ambulatory or ambulatory with aide
* Have a caregiver willing to accompany the patient to each visit, accept responsibility for supervising treatment and provided input to clinical outcome assessments
* Reside at home
* Speak English
* Amyloid positive PET-scan
* If they are on AD medications they must be stable on AD medications for at least three months prior to baseline
* Subjects ore willing/able to provide informed consent.

Exclusion Criteria:

* Patients with significant neurological disorder other than AD including hypoxia, stroke, traumatic brain injury
* A current psychiatric disorder according the DSM-IV diagnosis of major depression unless successfully treated on a stable dose of an antidepressant for at least 4 weeks and continues on stable dose throughout the study
* Any other DSM-IV Axis l diagnosis including other primary neurodegenerative dementia schizophrenia or bipolar depression
* A current diagnosis of uncontrolled diabetes mellitus (glucose values > 200 mg/ml).
* Patients with uncontrolled diabetes will be excluded because high glucose will alter the FDG-PET studies. The clinic that does PET (Columbia University Medical Center) excludes patients if glucose values exceed 200 mg/ml.
* A current diagnosis of active, uncontrolled seizure disorder
* A current diagnosis of probable or possible vascular dementia according to NINDS-AIREN
* An investigational drug during the previous 4 weeks
* A current diagnosis of severe unstable cardiovascular disease
* A current diagnosis of acute severe, or unstable asthmatic condition (e.g., severe chronic obstructive pulmonary disease (COPD),
* A current diagnosis of cardiac, renal or hepatic disease
* History of alcoholism, current or within past 5 years
* A disability that may prevent the patient from completing all study requirements (e.g., blindness, deafness, severe language difficulty)
* A1C less than or equal to 8
* Current diagnosis of cancer/active treatments

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Gibson, Ph.D., Principal Investigator — Burke Medical Research Institute; Pasquale Fonzetti, MD, PhD, Principal Investigator — Burke Rehabilitation Hospital
Locations (1):
- Burke, White Plains, New York, United States

REFERENCES:
- [Result] Gibson GE, Luchsinger JA, Cirio R, Chen H, Franchino-Elder J, Hirsch JA, Bettendorff L, Chen Z, Flowers SA, Gerber LM, Grandville T, Schupf N, Xu H, Stern Y, Habeck C, Jordan B, Fonzetti P. Benfotiamine and Cognitive Decline in Alzheimer's Disease: Results of a Randomized Placebo-Controlled Phase IIa Clinical Trial. J Alzheimers Dis. 2020;78(3):989-1010. doi: 10.3233/JAD-200896. PMID 33074237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from the Memory Evaluation and Treatment Service at the Burke Rehabilitation Center.
Groups:
- Benfotiamine: The patients in this arm will be treated with benfotiamine Benfotiamine: • To test whether increasing brain thiamine by administering 600 mg per day (300 mg/morning and 300 mg/evening) of benfotiamine for one year can slow cognitive decline in these patients as measured with the Alzheimer's Disease Assessment Scale (ADAS-COG).
  • To determine whether increasing brain thiamine availability with 600 mg (300 mg/morning and 300 mg/evening) per day of benfotiamine for one year can slow the decline in brain glucose metabolism in these patients as measured with Fluorodeoxyglucose Positron Emission Tomography(FGPET) in the posterior cingulate.
- Placebo: The patients in this arm will be treated with placebo
  To test whether increasing brain thiamine by administering 600 mg per day (300 mg/morning and 300 mg/evening) of benfotiamine for one year can slow cognitive decline in these patients as measured with the Alzheimer's Disease Assessment Scale (ADAS-COG).
  • To determine whether increasing brain thiamine availability with 600 mg (300 mg/morning and 300 mg/evening) per day of benfotiamine for one year can slow the decline in brain glucose metabolism in these patients. Placebo group received identical capsules without benfotiamine
Period: Overall Study
Arm/Group | Benfotiamine | Placebo
Started | 34 | 37
Completed | 30 | 33
Not Completed | 4 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 subject on the placebo arm was excluded from analysis due to taking benfotiamine from a commercial vendor.
Groups:
- Placebo: The patients in this arm will be treated with placebo
  Benfotiamine: • To test whether increasing brain thiamine by administering 600 mg per day (300 mg/morning and 300 mg/evening) of benfotiamine for one year can slow cognitive decline in these patients as measured with the Alzheimer's Disease Assessment Scale (ADAS-COG).
  • To determine whether increasing brain thiamine availability with 600 mg (300 mg/morning and 300 mg/evening) per day of benfotiamine for one year can slow the decline in brain glucose metabolism in these patients as measured with Fluorodeoxyglucose Positron Emission Tomography(FGPET) in the posterior cingulate.
- Total: Total of all reporting groups
Arm/Group | Benfotiamine | Placebo | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.74 (6.91) | 75.81 (7.19) | 75.77 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 11 | 18 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 33 | 35 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — All measures were made at patient interviews at the Burke Rehabilitation Hospital
  Participants
    United States | 34 | 36 | 70
MMSE Scores [Mean (Standard Deviation); unit: scores on a scale] — The Mini Mental State Examination (MMSE) is a set of standardized questions used to evaluate possible cognitive impairment and help stage the severity level of this impairment. Total scores on the MMSE range from 0 to 30. A total score of 0 indicates severe impairment, whereas a total score of 30 is normal. Scores of 20 to 25 are consistent with mild Alzheimer's Disease.
  scores on a scale | 25.32 (2.78) | 25.33 (2.52) | 25.33 (2.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ADAS-Cog Score
Description: The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) is a brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia. It is one of the most widely used cognitive scales in clinical trials and is considered to be the "gold standard" for assessing antidementia treatments. The ADAS-Cog range from 0 to 70, where higher scores indicate greater cognitive dysfunction.
Time Frame: Baseline, 1 year
Population: 1 subject on the placebo arm was excluded from analysis due to taking benfotiamine from a commercial vendor.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benfotiamine | Placebo
Number analyzed (Participants) | 34 | 36
score on a scale | 1.39 (5.63) | 3.26 (5.52)
Statistical Analysis 1: Comparison: Benfotiamine vs Placebo; Power was calculated based on expected difference in change on the ADAS-Cog of 3 points between the treatment and control groups. Estimates based on using a two-sided alpha of 0.05 and a standard deviation of 4, enrolling 29 patients per group, (N = 58) suggest 80% power to detect a mean change of 3 between treatment and placebo; Test type: Other; p = 0.125, t-test, 2 sided — Univariable (unadjusted) and a priori threshold for statistical significance is 0.05; Equal variance t-test; Mean Difference (Net) = 1.8691, Standard Deviation 5.5727

2. Secondary Outcome: Change From Baseline in Brain Glucose Utilization
Description: The AAL (Automatic Anatomical Labeling) atlas provides the taxonomy for 116 regions of interest, 90 of which capture non-cerebellar cortical regions. Signal averages from 9 cerebellar regions from each hemisphere were further averaged into one composite cerebellar region for each hemisphere, 'Cerebellum_L' and 'Cerebellum_R', which were comprised of the respective laterality averages of the regions: 'Cerebellum_Crus1 ' 'Cerebellum_Crus2 'Cerebellum_3' 'Cerebellum_4_5' 'Cerebellum_6' 'Cerebellum_7b' 'Cerebellum_8' 'Cerebellum_9' 'Cerebellum_10 '. Subsequently, these two composite regions are further combined with the bilateral paracentral lobules to provide one final composite for reference scaling. Concretely, the values from 'Cerebellum_L', 'Cerebellum_R', 'Paracentral_Lobule_L', and 'Paracentra_Lobule_R' were averaged. This final composite will serve as the denominator for the scaling operation of any ROI value prior to group-level analysis.
Time Frame: Baseline, 1 year
Population: 1 subject on the placebo arm was excluded from analysis due to taking benfotiamine from a commercial vendor.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Benfotiamine | Placebo
Number analyzed (Participants) | 34 | 36
ratio | -0.02 (0.02) | -0.01 (0.002)
Statistical Analysis 1: Comparison: Benfotiamine vs Placebo; Test type: Other — Univariable (unadjusted) and a priori threshold for statistical significance is 0.05; p = 0.7529, t-test, 2 sided; Equal variance t-test; Mean Difference (Net) = -0.00184, Standard Deviation 0.0225

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Score
Description: Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) is a caregiver-based Activities of Daily Living (ADL) scale composed of 23 items developed for use in dementia clinical studies. It was designed to assess the patient's performance of both basic and instrumental activities of daily living such as those necessary for personal care, communicating and interacting with other people, maintaining a household, conducting hobbies and interests, as well as making judgments and decisions. The range for the total ADCS-ADL score is 0 to 78. Higher scores equate with higher functioning.
Time Frame: Baseline, 1 year
Population: 1 subject on the placebo arm was excluded from analysis due to taking benfotiamine from a commercial vendor.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Benfotiamine: Patients were treated with 600 mg/day of benfotiamine
Arm/Group | Benfotiamine | Placebo
Number analyzed (Participants) | 34 | 36
score on a scale | -1.931 (0.9028) | -3.16129 (0.9816)
Statistical Analysis 1: Comparison: Benfotiamine vs Placebo; Test type: Other — Univariable (unadjusted) and a priori threshold for statistical significance is 0.05; p = 0.3687, t-test, 2 sided; Equal variance t-test; Mean Difference (Net) = -1.0636, Standard Deviation 4.8176

4. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Score
Description: The NPI assesses a wide range of behaviors encountered in dementia patients to provide a means of distinguishing frequency and severity of behavioral changes. Ten behavioral and two neuro-vegetative domains are evaluated through an interview with the caregiver. The total score ranges from 0 to 144. Higher scores suggest greater psychiatric impairment.
Time Frame: Baseline, 1 year
Population: 1 subject on the placebo arm was excluded from analysis due to taking benfotiamine from a commercial vendor.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benfotiamine | Placebo
Number analyzed (Participants) | 34 | 36
score on a scale | 6.69 (2.29) | 9.23 (3.8)
Statistical Analysis 1: Comparison: Benfotiamine vs Placebo; Test type: Other; p = 0.4850, t-test, 2 sided; Equal variance t-test; Mean Difference (Net) = 1.8203, Standard Deviation 13.8988

5. Secondary Outcome: Change From Baseline in Clinical Dementia Rating (CDR) Score
Description: The CDR was developed primarily for use in persons with dementia of the Alzheimer type (the equivalent of probable Alzheimer's Disease) and can also be used to stage dementia in other illnesses as well. The scores for the multiple items are summarized in one score. The CDR examines 6 categories of cognitive functioning domains. Each domain is scored on a scale ranging from 0 to 3 (including 0.5). A CDR-SB was generated as the sum of the values in each of the 6 domains. The CDR-SB sum scores range from 0 to 18, with higher scores indicating greater cognitive impairment and a 1 point worsening is considered a clinically significant symptom change.
Time Frame: Baseline, 1 year
Population: 1 subject on the placebo arm was excluded from analysis due to taking benfotiamine from a commercial vendor.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benfotiamine | Placebo
Number analyzed (Participants) | 34 | 36
score on a scale | 0.05 (0.08) | 0.22 (0.06)
Statistical Analysis 1: Comparison: Benfotiamine vs Placebo; Test type: Other; p = 0.0337, t-test, 2 sided — The a priori threshold for statistical significance is 0.05; Equal variance t-test; Mean Difference (Net) = 0.1907, Standard Deviation 0.3097

6. Secondary Outcome: Change From Baseline in Buschke Selective Reminding Test (SRT) Score
Description: The SRT is a standard diagnostic tool in the assessment of verbal memory. The Buschke SRT immediate total scores are compared between treated (benfotiamine) and control (placebo) groups. The immediate total score is the sum of correct responses over the 6 learning trials with scores ranging from 0 to 72. A score of 0 means severe impairment in memory. A score of 72 means there is no impairment in memory. For the purpose of determining effect over several trials between groups, the fractional change from the baseline of each group is compared.
Time Frame: Baseline, 1 year
Population: 1 subject on the placebo arm was excluded from analysis due to taking benfotiamine from a commercial vendor.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benfotiamine | Placebo
Number analyzed (Participants) | 34 | 36
score on a scale | 0.86 (1.1) | -1.12 (1)
Statistical Analysis 1: Comparison: Benfotiamine vs Placebo; Test type: Other — Univariable (unadjusted) and a priori threshold for statistical significance is 0.05; p = 0.315, t-test, 2 sided; Equal variance t-test; Mean Difference (Net) = -1.6161, Standard Deviation 5.6812

ADVERSE EVENTS:
Time Frame: 1 year
Description: 1 subject on the placebo arm was excluded from analysis due to taking benfotiamine from a commercial vendor.
Groups:
- Benfotiamine: To test whether increasing brain thiamine by administering 600 mg per day (300 mg/morning and 300 mg/evening) of benfotiamine for one year can slow cognitive decline in these patients as measured with the Alzheimer's Disease Assessment Scale (ADAS-COG).
  • To determine whether increasing brain thiamine availability with 600 mg (300 mg/morning and 300 mg/evening) per day of benfotiamine for one year can slow the decline in brain glucose metabolism in these patients. Placebo group received identical capsules without benfotiamine
Arm/Group | Benfotiamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 3/34 | 3/36
Other Adverse Events (participants affected / at risk) | 25/34 | 23/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Benfotiamine (N=34) | Placebo (N=36)
Surgery (General disorders) | 1 | 3
Stroke (General disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Benfotiamine (N=34) | Placebo (N=36)
Anxiety (Psychiatric disorders) | 5 | 4
Bruise (Skin and subcutaneous tissue disorders) | 2 | 5
Cold Symptoms (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Depression (Psychiatric disorders) | 1 | 2
Dizziness (Ear and labyrinth disorders) | 3 | 3
Fall (Injury, poisoning and procedural complications) | 6 | 12
Head Injury (Injury, poisoning and procedural complications) | 0 | 2
Heart Arrhythmia (Cardiac disorders) | 1 | 2
Pain (Nervous system disorders) | 5 | 4
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sprain (Injury, poisoning and procedural complications) | 0 | 2
Allergy (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT02292238/Prot_SAP_000.pdf